CLINICAL TRIAL: NCT00810758
Title: A Phase 1, Randomized, Placebo Controlled, Blinded (3rd Party Open), Sequential, Multiple-Dose Escalation Study To Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PF-04878691 In Healthy Volunteers
Brief Title: Multiple Oral Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PF-04878691
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: B1201002
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Hepatitis C Virus
Keywords: HCV; Toll-like receptor 7; Multiple oral dose escalation study of PF-04878691
MeSH Terms: conditions — Hepatitis C | interventions — N-(4-(4-amino-2-ethyl-1H-imidazo(4,5c)quinolin-1-yl)butyl)methanesulfonamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-04878691 (Experimental)
  Interventions: Drug: PF-04878691 3mg; Drug: PF-04878691 6mg; Drug: PF-04878691 9mg

INTERVENTIONS:
Drug: PF-04878691 3mg — Oral solution, 3mg, twice weekly, 2 weeks
Drug: PF-04878691 6mg — Oral solution, 6mg, twice weekly, 2 weeks
Drug: PF-04878691 9mg — Oral solution, 9mg, twice weekly, 2 weeks

SUMMARY:
To assess the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple oral doses of PF-04878691.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18-55, inclusive.
* Body Mass Index (BMI) of 18-30 kg/m2; total body weight >50kg (110lbs).

Exclusion Criteria:

* Pregnant or nursing females.
* Females of child-bearing potential.
* Evidence of history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, allergic or autoimmune disease or clinical findings at screening.
* Smoking within the previous 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety and toleration of multiple ascending oral doses of PF-04878691 | 3 weeks

SECONDARY OUTCOMES:
To assess the pharmacokinetics and pharmacodynamics with regards to specific biomarkers of immune stimulation of PF-04878691 | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1201002&StudyName=Multiple%20Oral%20Dose%20Study%20to%20Evaluate%20the%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20and%20Pharmacodynamics%20of%20PF-04878691